CLINICAL TRIAL: NCT06235294
Title: Effects of Resveratrol Supplementation on Oocyte Quality in Advanced Maternal Aged Women Undergoing in Vitro Fertilization.
Brief Title: Effects of Resveratrol Supplementation on Oocyte Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA-01-23
Record Dates: First submitted 2024-01-14; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Aging; Infertility
Keywords: in vitro fertilization; oocyte quality; resveratrol
MeSH Terms: conditions — Infertility | interventions — Resveratrol; Folic Acid

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to groups according to random numbers generated by a computer and implemented via a sealed envelope. The random allocation, enrollment of patients and assignment of intervention will be performed by the principal investigator.
Who Masked: Participant, Care Provider
Masking Description: Patients, physicians, and embryologists will be blinded to group assignments of the participants in the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Experimental): Daily capsule of 200 mg Polygonum cuspidatum yielding 100 mg/day resveratrol (trans-3,5,4'-trihydroxystilbene)
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator): Daily capsule of 400 mcg folic acid.
  Interventions: Dietary Supplement: Folic acid

INTERVENTIONS:
Dietary Supplement: Resveratrol — Daily capsule of 200 mg Polygonum cuspidatum (Solgar®, Dietimport, Lisboa, Portugal) yielding 100 mg/day resveratrol (trans-3,5,4'-trihydroxystilbene), by morning, every day during the 3 months preceding in vitro fertilization treatment.
  Arms: Resveratrol
Dietary Supplement: Folic acid — Daily capsule of 400 mcg folic acid (Solgar®, Dietimport, Lisboa, Portugal), by morning, every day during the 3 months preceding in vitro fertilization treatment.
  Arms: Placebo

SUMMARY:
The goal of this randomized, double-blind, placebo-controlled clinical trial is to verify if 3-month oral supplementation with resveratrol can enhance the oocyte quality in advanced maternal age women undergoing in vitro fertilization (IVF).

Participants will take a daily capsule of resveratrol or placebo during the 3 months preceding their IVF treatment. They will then follow the same treatment protocol as non-participant patients.

DETAILED DESCRIPTION:
The study will be conducted in the Reproductive Medicine Unit of an Academic Hospital.

Eligible participants who meet the inclusion and exclusion criteria will be randomly assigned to one of the following groups:

1. Resveratrol (study group) or
2. Placebo (control group).

Supplementation

Women in the study group will take a daily capsule of 200 mg Polygonum cuspidatum (Solgar®, Dietimport, Lisboa, Portugal) yielding 100 mg/day resveratrol (trans-3,5,4'-trihydroxystilbene). Women from control group will take a daily capsule of 400 mcg folic acid (Solgar®, Dietimport, Lisboa, Portugal), a vitamin widely prescribed to women who intend to achieve pregnancy for prevention of neural tube defects). Participants will be instructed to take the capsules by morning, every day during the 3 months preceding their IVF treatment. Oral intake of resveratrol/placebo will be discontinued after oocyte retrieval due to the potential adverse effects of resveratrol on endometrial decidualization. Package of resveratrol and placebo will be identical. Compliance of the participant to the intervention will be measured using capsule count. Participants will be asked to keep their usual lifestyle including nutrition and physical activity level.

Ovarian stimulation

GnRH antagonist protocol will be used in all the patients. On day 2 or 3 of the menstrual cycle, daily subcutaneous (SC) injections of rFSH are given up to the day of human chorionic gonadotropin (hCG) administration, when at least three leading follicles reached a mean diameter of 17 mm. Doses of rFSH range from 150 to 300 IU/day depending on the women's age, body mass index (BMI), AFC and AMH. Administration of a daily dose of 0.25 mg of gonadotropin releasing hormone antagonist (GnRHa) (Cetrotide ®, Merck, Netherlands; or Orgalutran ®, Organon, Netherlands) is initiated when the larger follicle reaches a mean diameter of 14 mm. Transvaginal oocyte retrieval is scheduled to 36 hours after choriogonadotropin alfa (α-hCG) administration. Luteal phase support with progesterone is initiated on the day of the oocyte retrieval with 200 mg of micronized intravaginal progesterone every 8 hours (Progeffik ®, EFIKK, France).

In vitro fertilization and embryo transfer

According to the couples's indication, IVF or ICSI is performed. Fertilization is assessed after 18 hours, and oocyte maturational stage is assessed and registered. Embryo cleavage is assessed every 24 hours. Embryo transfer is performed 5 days after oocyte retrieval under ultrasound guidance. All remaining good quality embryos will be vitrified and transferred in subsequent menstrual cycles. If fresh transfer is canceled for clinical reasons, frozen embryo transfer will also be scheduled. Before frozen embryo transfer, patients will start exogenous hormone therapy for endometrial preparation. This therapy is initiated on day 1 of menstrual cycle and consists of 150 mcg of estradiol transdermal patches (Dermestril®, BGP, Lisboa, Portugal) replaced every 3 days. On day 12-14, a pelvic ultrasound is performed to assess endometrial development. If the endometrial thickness is > 7 mm, 400 mg vaginal micronized progesterone (Cyclogest®, Gedeon Richter, Budapest, Hungria) twice daily was added to the treatment scheme. Fourteen days after oocyte retrieval a quantitative serum value of β-hCG is obtained and a transvaginal ultrasound is scheduled one week later in case of a positive result (biochemical pregnancy). Clinical pregnancy is established by the ultrasonography visualization of a gestational sac. Ongoing pregnancy was defined by a viable intrauterine pregnancy of at least 12 weeks duration confirmed on an ultrasound scan. The outcomes of fresh and vitrified-warmed embryo transfer will be analyzed. Live birth was defined as the delivery of one or more live babies. Miscarriage was defined by a spontaneous pregnancy termination before the gestational age of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women with infertility undergoing IVF/ICSI
* Ovarian stimulation with GnRH-antagonist protocol
* Age 35-40 years old

Exclusion Criteria:

* Severe male factor (oligospermia or azoospermia)
* Low ovarian reserve (AMH < 1.1. ng/mL)
* Poor response to ovarian stimulation (< 3 oocytes)
* Polycystic ovarian syndrome (Rotterdam criteria)
* Ovarian endometriosis (endometrioma > 30 mm)
* Uterine anomalies (congenital or acquired)
* Diabetes Mellitus
* Concurrent use of any vitamin (except folic acid)

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of good-quality embryos | 4 months
  Embryos available to transfer or cryopreservation.

SECONDARY OUTCOMES:
Number of oocytes and mature oocytes | 4 months
  Total oocytes and metaphase-II oocytes retrieved.
Fertilization rate | 4 months
  Percentage of oocytes with two pronuclei by the number of COCs retrieved)
Cleavage rate | 4 months
  Percentage of 2-cell stage embryos by the number of COCs retrieved
Biochemical pregnancy rate | up to 15 months
  Percentage of positive B-hCG in serum by initiated cycle
Clinical pregnancy rate per cycle | up to 15 months
  Proportion of positive clinical pregnancies by initiated cycle
Clinical pregnancy rate per embryo transfer | up to 15 months
  Proportion of positive clinical pregnancies by embryo transfer
Ongoing pregnancy rate | up to 15 months
  Proportion of ongoing pregnancies (viable intrauterine pregnancy of at least 12 weeks)
Cumulate live birth rate | up to 15 months
  Number of deliveries with at least one live birth resulting from one initiated cycle